CLINICAL TRIAL: NCT01272830
Title: A Prospective Double-Blinded Clinical Trial Using Apatone®B for Care and Treatment of Proven Non-Infected Symptomatic Postoperative Total Joint Arthroplasties
Brief Title: Double-Blinded Clinical Trial Using Apatone®B for Symptomatic Postoperative Total Joint Replacements
Acronym: Apatone-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IC-MedTech Corporation (Industry)
Collaborators: Summa Health System (Other); Crystal Clinic Orthopaedic Center LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Summa-09136
Record Dates: First submitted 2010-12-17; First posted 2011-01-10 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2017-10

CONDITIONS: Edematous; Synovitis; Foreign Body Reaction; Osteolysis
Keywords: total joint arthroplasty; synovitis; ALVAL (Aseptic Lymphocyte-Dominant Vasculitis-Associated Lesion); osteolysis; periprosthetic metallosis
MeSH Terms: conditions — Edema; Synovitis; Foreign-Body Reaction; Osteolysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral Apatone®B (Experimental): An amalgam of Vitamins C & K3
  Interventions: Drug: Apatone®B
- Placebo (Placebo Comparator): Oral capsule of similar appearance and taste without Apatone®B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Two capsules taken twice daily with meals
  Arms: Placebo
Drug: Apatone®B — Two capsules taken twice daily with meals
  Arms: oral Apatone®B

SUMMARY:
This research study is being conducted to determine if taking oral (by mouth in pill form) Apatone®B (a combination of Vitamins C and K3) will reduce chronic joint discomfort and improve function of non-infected symptomatic postoperative total joint replacements.

DETAILED DESCRIPTION:
To perform a prospective, randomized, double-blind clinical trial to determine if oral Apatone®B, an amalgam of vitamins C and K3, has a therapeutic efficacy beyond the conservative care customarily used to reduce inflammatory synovitis and to increase the functional capacity of proven non-infected symptomatic postoperative total joint replacements.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative Total joint replacement with osteoarthritis as the underlying pathology
* Proven non-infected symptomatic Total Joint Arthroplasty (TJA) (joint implanted for >12 months post-op)
* Age (50 to 85 years of age); based on a 10% trim of the age distribution for Summa Health System TJAs (7/1/08-6/30/2009).

Exclusion Criteria:

* An infection of any kind (prior to, or during the study)
* Rheumatoid arthritis as the underlying pathology
* Cortisone injection received <6 months prior to study enrollment
* Insulin dependent diabetes
* Diagnosed immunodeficiency
* On dialysis or have poor kidney function
* Anti-coagulant medication (e.g., Coumadin or >100mg of Aspirin daily)
* Anti-seizure medication (e.g., Dilantin)
* Steroidal medication (e.g., Prednisone, Advair or Symbicort)
* NSAIDS (e.g., Celebrex or Toradol); a 14-day washout period will be allowed
* bisphosphonates (e.g., Fosamax, Actonel, Aredia, Didronel, Boniva or Reclast)
* hormonal therapy (e.g., Estrogen, Progesterone or Testosterone)
* Cancer (active or in remission)
* Planned concurrent vitamins exceeding a standard daily multivitamin or exceeding the Recommended Daily Allowance (RDA) for individual vitamins if used alone; a 72 hour wash out period will be allowed
* A glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Pregnant or lactating; females who are in their reproductive years must have a negative serum pregnancy
* Lactose intolerant
* Citric acid intolerant

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Bear, MD, Principal Investigator — Crystal Clinic Orthopaedic Center LLC; Mark W Kovacik, BS, Study Director — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 57 subjects were consented to participate.
Pre-assignment Details: Following consenting, 6 subjects did not meet the study inclusion/exclusion criteria, thus never received the study drug.
  1 - Abnormal Liver Panel: very low Hemoglobin/Hematocrit levels
  1 - Glucose-6-phosphate dehydrogenase (G6PD) deficiency
  3 - X-rays revealed loose or mal-positioned component(s)
  1 - Prescribed steroids prior to study drug
Period: Overall Study
Arm/Group | Oral Apatone®B | Placebo
Started | 25 | 26
Completed | 17 | 21
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Apatone®B | Placebo | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.5) | 65.4 (9.6) | 63.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 8 | 9 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 21 | 38
Weight [Mean (Standard Deviation); unit: kilograms] | 96.7 (20.4) | 100 (16.8) | 99 (18.5)
Height [Mean (Standard Deviation); unit: centimeters] | 171.7 (9.9) | 169.8 (8.6) | 170.6 (9.2)
Time elapsed since TKA [Mean (Standard Deviation); unit: years] — TKA - Total Knee Arthroplasty
  years | 2.5 (1.9) | 4.0 (3.3) | 3.3 (2.9)
Initial Pain Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — VAS Scale range (0-100 )
  Higher VAS score indicate worst knee pain.
  units on a scale | 57 (24.1) | 46.8 (24.9) | 51.4 (25.1)

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analog Scale (VAS)
Description: Pain Visual Analog Scale (VAS)
  Scale range (0-100) A higher VAS score indicate worse knee pain
Time Frame: 13-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Apatone®B | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale
  Baseline | 57 (24.1) | 46.8 (24.9)
  13 Weeks | 39.7 (27.4) | 39.1 (29.1)
Statistical Analysis 1: Comparison: Oral Apatone®B; Change from baseline data; Test type: Superiority; p = 0.0063, paired t-test — Significance threshold p<0.05
Statistical Analysis 2: Comparison: Placebo; Changes from baseline data; Test type: Superiority; p > 0.05, paired t-test — Significant threshold p<0.05

2. Secondary Outcome: Surrogate Endpoint Markers (SEBs)
Description: HSS = Hospital for Special Surgery Knee Score , KSS = Knee Society Knee Score.
  * Scale range HSS total: 100-90 Excellent; 80-89 Very Good; 70-79 Good; 60-69 Fair; below 60 Poor
  * Scale range HSS pain walking: No Pain 15; Mild Pain 10; Moderate Pain 5; Severe Pain 0 (**this is an element of the HSS total)
  * Scale range KSS: 80-100 Excellent; 70-79 Good; 60-69 Fair; below 60 Poor
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Apatone®B | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale
  HSS Pain Walking- Baseline | 5.9 (5.4) | 6.9 (4.3)
  HSS Pain Walking-13 Weeks | 9.1 (6.2) | 7.9 (4.4)
  HSS Total-Baseline | 69.6 (14.3) | 71.9 (11.6)
  HSS Total-13 Weeks | 76.6 (16.7) | 74.5 (11.1)
  KSS Total Pain-Baseline | 56.2 (19.4) | 59.0 (14.0)
  KSS Total Pain-13 Week | 65.3 (20.1) | 63.0 (18.4)
Statistical Analysis 1: Comparison: Oral Apatone®B; Change from baseline data (HSS pain walking); Test type: Superiority; p = 0.0226, paired — Significance threshold p<0.5
Statistical Analysis 2: Comparison: Oral Apatone®B; Change from baseline data (HSS total score); Test type: Superiority; p = 0.0375, paired t-test — Significance threshold P<0.05
Statistical Analysis 3: Comparison: Oral Apatone®B; Change from baseline data (KSS knee pain); Test type: Superiority; p = 0.0391, paired t-test — Significance threshold p<0.05
Statistical Analysis 4: Comparison: Placebo; Changes from baseline data (HSS pain walking); Test type: Superiority; p = 0.2137, paired t-test
Statistical Analysis 5: Comparison: Placebo; Change from baseline data (HSS total score); Test type: Superiority; p = 0.1312, paired t-test
Statistical Analysis 6: Comparison: Placebo; Change from baseline data (KSS knee pain); Test type: Superiority; p = 0.1578, paired t-test

3. Secondary Outcome: TGFBeta Levels
Description: The final synovial aspirates obtained from the symptomatic knee of each subject were analyzed using Quantikine and Pyrilinks-D enzyme-linked immunosorbent assay kits from R&D Systems (Minneapolis, MN) and Metra Biosystems (Mountain View, CA), respectively.
  Lower TGFBeta concentrations represent a better outcome.
Time Frame: Baseline and 13 Weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Oral Apatone®B | Placebo
Number analyzed (Participants) | 17 | 21
pg/mL
  Baseline | 3197.4 (2793.5) | 2089.2 (2879.7)
  13 Weeks | 2572.2 (2879.7) | 1572.2 (1803.9)
Statistical Analysis 1: Comparison: Oral Apatone®B; Changes from baseline data; Test type: Superiority; p = 0.0083, t-test — Significance threshold p<0.05
Statistical Analysis 2: Comparison: Placebo; Change from baseline data; Test type: Superiority; p > 0.05, paired t-test — Significant threshold p<0.05

4. Secondary Outcome: Deoxypyridinoline Levels
Description: The final synovial aspirates obtained from the symptomatic knee of each subject were analyzed using Quantikine and Pyrlinks-D enzyme-linked immunosorbent assay kits from R&D Systems(minneapolis, MN) and Metra Biosystems (Mountain View, CA) respectively.
  Lower DPD concentrations represent a better outcome
Time Frame: Baseline and 13 Weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Oral Apatone®B | Placebo
Number analyzed (Participants) | 17 | 21
nmol/L
  Basline | 8.0 (6.0) | 5.9 (1.3)
  13 Weeks | 6.4 (1.5) | 6.1 (1.8)
Statistical Analysis 1: Comparison: Oral Apatone®B; Change from baseline data; Test type: Superiority; p = 0.01, ANOVA — Significance threshold p<0.05
Statistical Analysis 2: Comparison: Placebo; Changes from baseline data; Test type: Superiority; p > 0.05, paired t-test; Significant threshold p<0.05

ADVERSE EVENTS:
Description: All adverse events (AEs) were classified by the investigator with respect to severity (mild, moderate, severe and potentially life threatening). No AEs classified as potentially life threatening were reported during the course of this study, nor were there any deaths.
Arm/Group | Oral Apatone®B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/21
Other Adverse Events (participants affected / at risk) | 14/17 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Apatone®B (N=17) | Placebo (N=21)
Knee pain - hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Outcome - not recovered, ongoing. Did not finish study; revision knee surgery elected before trial completion.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Apatone®B (N=17) | Placebo (N=21)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Knee discomfort left and right (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Entire body ached (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Extreme knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall outdoors, hit head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Painful knee aspiration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulled muscle right knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Right calf pain, possible blood clot (Vascular disorders) | 1 (1) | 0 (0)
Right knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Slipped on ice; cracked rib (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Swelling of knees (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
13th week elevated PT, PTT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Knee discomfort right (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee pain left (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Repeated PT, PTT one week later (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
limited accrual due to meeting stringent study inclusion/exclusion criteria.Stringent inclusion/exclusion created to allow SEB analyses w/o interference or artifacts,& not due to study drug issues,interaction or limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Published articles to be reviewed/approved by IC-MedTech prior to publication.